CLINICAL TRIAL: NCT00701792
Title: Randomized Trial Comparing Liver Transplantation to Alternative Therapies for Patients With Pugh B Alcoholic Cirrhosis
Brief Title: Liver Transplantation Versus Alternative Therapies for Patients With Pugh B Alcoholic Cirrhosis
Acronym: TRANSCIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: M. FLAMMARION - Directeur des Projets, de la Recherche CLinique et de l'Innovation, Centre Hospitalier Universitaire de Besancon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N/1993/04
Record Dates: First submitted 2008-06-05; First posted 2008-06-19 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Cirrhosis
Keywords: cirrhosis transplantation
MeSH Terms: conditions — Fibrosis | interventions — Liver Transplantation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): surgery : liver transplantation
  Interventions: Procedure: liver transplantation
- 2 (Active Comparator): standard care for liver disease
  Interventions: Other: standard care for liver disease

INTERVENTIONS:
Procedure: liver transplantation — liver transplantation
  Arms: 1
Other: standard care for liver disease — standard care for liver disease included therapy for ascitis (spironolactone, furosemide), portal hypertension (oesophageal varices ; propranolol), encephalopathy (lactulose), and bacterial infections whatever their localization (prophylaxis of spontaneous peritonitis with norfloxacin). All medical or instrumental procedures were allowed. Patients undergoing iterative paracentesis, variceal band ligation or sclerotherapy, peritoneojugular shunt (LeVeen), transjugular intrahepatic portosystemic shunt (TIPS) or surgical portocaval anastomosis were considered as receiving "standard medical therapy".
  Arms: 2

SUMMARY:
Liver transplantation has been universally recognized to improve survival of patients suffering from end-stage (Pugh C) alcoholic cirrhosis. However, for Pugh B patients, the benefit of liver transplantation remains to be demonstrated. The aim of the present study was to compare the outcome of Pugh B patients with alcoholic cirrhosis randomly assigned for immediate liver transplantation (group 1) or standard treatments (group 2).

DETAILED DESCRIPTION:
120 patients (60 per group) were included. The therapeutic strategy defined by randomization was achieved in 68% of group 1 patients and 75% of group 2 patients (NS). All-causes death and cirrhosis-related death were not different in group 1 and group 2 patients: the five-year survival rate was 58% in group 1 and 69% in group 2 patients (NS). Through multivariate analysis, the independent predictors of long-term survival were absence of ongoing alcohol consumption (p<0.001), recovery from Pugh C (p=0.046), and baseline Pugh score<8 (p=0.029). Liver transplantation was associated with a higher rate of de novo malignancies (30.4% vs. 7.8%, OR=5.1, p=0.001).

ELIGIBILITY:
Inclusion Criteria:

* cirrhosis
* age 18-65yrs
* Pugh B
* written consent

Exclusion Criteria:

* HIV, HBV or HCV infection
* hepatocellular carcinoma
* Pugh A or Pugh C cirrhosis
* creatinin >200µMol/L
* sepsis
* psychiatric disorders
* extrahepatic neoplasia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1994-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
all causes mortality | five years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Phillipe MIGUET, Study Chair — Service d'Hépatologie - CHU de Besançon
Locations (13):
- France (13):
  - service d'hépatologie CHU jean Minjoz, Besançon
  - CHRU CAEN - Service d'hépato-gastroentérologie, Caen
  - Hôpital Beaujon - Hépato-gastroentérologie, Clichy
  - CHU Henri Mondor - Hépato-gastroentérologie, Créteil
  - Hépato-gastroenterologie CHU Bocage, Dijon
  - Centre d'épidémiologie de population EPI 106, Dijon
  - Hôpital Bon secours - Hépato-gastroentérologie, Metz
  - Hôpital Saint-Eloi - Hépato-gastroentérologie, Montpellier
  - Hôpital Pitié-Salpétrière - Hépato-gastroentérologie, Paris
  - Hepato-gastroenterologie, Poitiers
  - CHU Reims - hépato-gestroentérologie, Reims
  - Clinique des maladies du foie Hôpital Pontchailloux, Rennes
  - Hôpital Purpan - Hépato-gastroentérologie, Toulouse

REFERENCES:
- [Derived] Vanlemmens C, Di Martino V, Milan C, Messner M, Minello A, Duvoux C, Poynard T, Perarnau JM, Piquet MA, Pageaux GP, Dharancy S, Silvain C, Hillaire S, Thiefin G, Vinel JP, Hillon P, Collin E, Mantion G, Miguet JP; TRANSCIAL Study Group. Immediate listing for liver transplantation versus standard care for Child-Pugh stage B alcoholic cirrhosis: a randomized trial. Ann Intern Med. 2009 Feb 3;150(3):153-61. doi: 10.7326/0003-4819-150-3-200902030-00004. PMID 19189904